CLINICAL TRIAL: NCT05418582
Title: A Phase 1, Single-Center, Nonrandomized, Open-Label, 2-Part, Fixed-Sequence, Drug-Drug Interaction Study to Assess the Pharmacokinetics of DZD9008 When Orally Administered Alone, When Coadministered With Itraconazole, and When Coadministered With Carbamazepine in Healthy Adult Subjects
Brief Title: Drug-drug Interactions Between DZD9008 and Itraconazole/Carbamazepine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: DZ2021E0008
Record Dates: First submitted 2022-05-28; First posted 2022-06-14 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Carbamazepine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DZD9008 and itraconazole (Experimental): Subjects in arm 1 will receive DZD9008 single dose on Day 1, and the second dose of DZD9008 along with itraconazole after the wash-out period.
  Interventions: Drug: DZD9008 and intraconazole
- DZD9008 and carbamazepine (Experimental): Subjects in arm 2 will receive DZD9008 single dose on Day 1, and the second dose of DZD9008 along with carbamazepine after the wash-out period.
  Interventions: Drug: DZD9008 and carbamazepine

INTERVENTIONS:
Drug: DZD9008 and intraconazole — All subjects will receive DZD9008 single dose on Day 1, and the second dose of DZD9008 along with itraconazole after the wash-out period.
  Arms: DZD9008 and itraconazole
Drug: DZD9008 and carbamazepine — All subjects will receive DZD9008 single dose on Day 1, and the second dose of DZD9008 along with carbamazepine after the wash-out period.
  Arms: DZD9008 and carbamazepine

SUMMARY:
This is a Phase 1, single-center, nonrandomized, open-label, 2-part, fixed-sequence, drug-drug interaction (DDI) study to assess the effect of multiple doses of itraconazole, a CYP3A4 enzyme inhibitor, on the single dose PK of DZD9008 in healthy adult subjects (Part A) and to assess the effect of multiple doses of carbamazepine, a CYP3A4 inducer, on the single dose PK of DZD9008 in healthy adult subjects (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aging 18 to 55 years with Body mass index (BMI) 18.0 to 30.0 kg/m2.
* Weight : ≥ 55 kg for males and ≥ 45 kg for females.
* Healthy status as defined by the absence of evidence of any clinically significant, in the opinion of the Investigator, active or chronic disease following a detailed medical and surgical history, a complete physical examination.
* Ability and willingness to abstain from alcohol-, caffeine-, and methylxanthine-containing beverages or food during the stay in study center.
* No clinically significant hematological or coagulation abnormalities, as judged by the Investigator.
* Male subjects and female subjects of childbearing potential must agree to use protocol-specified method(s) of contraception and comply with pregnancy precautions.
* All nonregular medication (including over-the-counter [OTC] medication, health supplements, and herbal remedies such as St. John's wort extract) must have been stopped at least 14 days or 5 half-lives, if known (whichever is longer) prior to the admission to the clinical research center.
* Normal baseline pulmonary function tests (≥ 80% predicted normal for spirometry, lung volumes).
* Normal baseline ECG (QTcF < 450 msec, PR < 220 msec).
* Adequate organ function including hepatic, renal, cardiac, and bone marrow function, as determined by the Investigator.

Exclusion Criteria:

* Employee of PRA or the Sponsor.
* Any condition which, in the opinion of the Investigator, would interfere with the subject's ability to provide informed consent, comply with study instructions, confound interpretation of study results, or endanger the subject if he or she takes part in the trial.
* Women who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 30 days after dosing of study drug.
* For all females of childbearing potential: positive pregnancy test at screening and at admission to the clinic.
* Males with female partners who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 90 days after dosing of study drug.
* Use of any investigational drug or device within 30 days of the first dose of study drug.
* Any disease which, in the opinion of the Investigator, poses an unacceptable risk to the subjects.
* Clinically relevant issues of visual function as determined from the medical history and physical exams, as judged by the Investigator.
* Clinically significant history of any drug sensitivity, drug allergy, or food allergy, as determined by the Investigator (such as anaphylaxis, hepatotoxicity, or treatment with steroids or epinephrine). Confirmatory circumstances would include treatment with epinephrine or in Emergency Department.
* History of allergy or hypersensitivity to DZD9008, or other drugs similar in class (EGFR/HER2/BTK inhibitor) or similar in chemical structure to DZD9008, as judged by the Investigator.
* History of major surgery or blood transfusion within 30 days prior to the first drug administration.
* History of malignancy of any type, except for the following: surgically excised non-melanomatous skin cancers more than 5 years prior to receiving the investigational medicinal product.
* Evidence of clinically significant or relevant renal, hematological, endocrine, pulmonary, GI, cardiovascular, hepatic, psychiatric, neurological, or allergic disease, as judged by the Investigator.
* Manifestation of malabsorption due to prior GI surgery, GI disease, or any other reason that may affect the absorption of DZD9008.
* Positive result from a COVID-19 test per local policy and requirement.
* Positive test result for alcohol and/or drugs of abuse at screening or on Day1.
* Positive test result from Quantiferon-TB Gold test.
* Presence of pulmonary infections or other clinically significant active infection within 30 days of informed consent.
* Received COVID-19 vaccine or any live vaccine within 4 weeks prior to the first dose of the investigational medicinal product.
* Self-reported substance abuse (eg, alcohol, licit, or illict drugs) within 12 months of screening.
* Using tobacco or nicotine products within 90 days prior to the first drug administration.
* Strenuous activity, sunbathing, and contact sports within 48 hours (2 days) prior to admission to the clinical facility through follow-up.
* History of donation of more than 500 mL of blood within 60 days prior to dosing in the clinical research center or planned donation before 30 days has elapsed since intake of study drug.
* Plasma or platelet donation within 7 days of dosing and through follow-up.
* History within the previous 12 months of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink=12 oz beer, 5 oz wine, and 1.5 oz spirits). Alcohol consumption will be prohibited 72 hours prior to admission to the clinical facility and until discharge in the last study period.
* Positive screening test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or HIV 1 and 2 antibodies.
* Consumption of any nutrients known to modulate CYP450 enzymes activity (eg, grapefruit or grapefruit juice, pomelo juice, star fruit, or Seville [blood] orange products) within 14 days prior to administration of study drug and during the study (until after discharge in the last study period).
* Abnormal echocardiogram (ECHO) at baseline (eg, left ventricular ejection fraction [LVEF] < 50%), as judged by the Investigator.
* History of allergy, severe adverse reaction, intolerance, or hypersensitivity to itraconazole or other azole antifungals, as determined by the Investigator. (Part A Only)
* History of allergy, severe adverse reaction, intolerance, or hypersensitivity to carbamazepine, carboxamide derivatives (eg, oxcarbazepine), or other drugs that are structurally-related to carbamazepine, which include, but are not limited to tricyclic antidepressants (eg, amitriptyline, desipramine, imipramine, protriptyline, or nortriptyline), as judged by the Investigator. (Part B Only)
* Individuals who have Asian ancestry (including those who have one or more Asian grandparents). (Part B Only)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of DZD9008 when dosed alone or coadministered with itraconazole (Part A） | up to 11 days after study drug administration
Time to reach maximum plasma concentration (tmax) of DZD9008 when dosed alone or coadministered with itraconazole (Part A) | up to 11 days after study drug administration
Area under the concentration-time curve from time 0 to time of last quantifiable concentration (AUC0-t) when dosed alone or coadministered with itraconazole (Part A) | up to 11 days after study drug administration
Area under the concentration-time curve from time 0 to infinity (AUC0-inf) when dosed alone or coadministered with itraconazole (Part A) | up to 11 days after study drug administration
Maximum plasma concentration (Cmax) of DZD9008 when dosed alone or coadministered with carbamazepine (Part B) | up to 10 days after study drug administration
Time to reach maximum plasma concentration (tmax) of DZD9008 when dosed alone or coadministered with carbamazepine (Part B) | up to 10 days after study drug administration
Area under the concentration-time curve from time 0 to time of last quantifiable concentration (AUC0-t) when dosed alone or coadministered with carbamazepine (Part B) | up to 10 days after study drug administration
Area under the concentration-time curve from time 0 to infinity (AUC0-inf) when dosed alone or coadministered with carbamazepine (Part B) | up to 10 days after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Tianwei Zhang, Study Director — Dizal Pharma
Locations (1):
- Pharmaceutical Research Associates, Inc., Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No